CLINICAL TRIAL: NCT06776952
Title: A Randomized, Double-blind, Multicenter Phase III Study of XNW5004 Tablets in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Evopoint Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XNW5004-III-01
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: XNW5004 ; Chidamide placebo
- Treatment group B (Experimental)
  Interventions: Drug: XNW5004 placebo; Chidamide

INTERVENTIONS:
Drug: XNW5004 ; Chidamide placebo — XNW5004 + Chidamide placebo
  Arms: Treatment group A
Drug: XNW5004 placebo; Chidamide — XNW5004 placebo + Chidamide
  Arms: Treatment group B

SUMMARY:
This is a randomized, double-blind, multi-center, phase III clinical trial designed to evaluate the efficacy of XNW5004 tablets versus Chidamide in Relapsed/Refractory PTCL, with a target of enrolling 120 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years (inclusive)，gender not limited.
* Pathologically diagnosed, relapsed or refractory peripheral T-cell lymphoma.
* Disease status defined as relapsed or refractory after >=1 prior systemic treatment lines, and have not received treatment with HDAC inhibitors, subjects with NK/T-cell lymphoma require treatment with a regimen containing asparaginase/protease, subjects with CD30 positive ALCL require prior treatment with Brentuximab vedotin.
* Subjects who have received prior radiotherapy are allowed to enroll, but radiotherapy alone is not considered a systemic therapy.
* Having at least one measurable lesion for evaluation.
* Agree to provide archived tumor tissue samples or fresh tumor tissue samples that meet the requirements.
* Life expectancy of at least 12 weeks.
* Subjects must have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Have adequate organ function.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to the first dose of study drug. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test is required.Non-sterile subjects must be willing to use a highly effective contraception (e.g., IUD, pill, or condom) for the duration of the study and for 6 months after the last dose of study drug unless their partner is sterilized. For male subjects whose partner is a woman of childbearing potential, surgical sterilization or agreement to use effective contraception for the duration of the study and for 6 months after the last dose of study drug is required. In addition, males must agree not to donate sperm during the study participation and for at least 6 months after the last dose of study drug.
* Able to provide written informed consent form prior to the commencement of any study activity/procedure.

Exclusion Criteria:

* Prior exposure to EZH2 inhibitor(s) or EZH1/2 inhibitor(s).
* Prior exposure to HDAC inhibitor(s).
* Subjects with known hypersensitivity to the study drug or its active ingredients or excipients.
* Subjects who have received anti-tumor therapy, such as chemotherapy, immunotherapy, radiotherapy, and targeted therapy, within 4 weeks or 5 half-lives (whichever is shorter) before the first dose of the study drug, received CAR-T therapy within 12 weeks prior to the first dose of the study drug, autologous hematopoietic stem cell transplantation (Auto-HSCT) within 3 months prior to the first dose of the study drug.
* Subjects who have received other anti-tumor investigational drug treatment within 28 days prior to the first dose of XNW5004 in this study.
* Subjects who have undergone major surgery within 4 weeks prior to the start of study treatment or who intend to undergo major surgery during this study (except for procedures such as puncture or lymph node biopsy).
* Subjects who have an allogeneic hematopoietic stem cell transplantation or solid organ transplantation.
* Subjects who have received systemic treatment with corticosteroids (prednisone at a dose of > 10 mg per day or equivalent doses of other glucocorticoids) or other immunosuppressive drugs within 14 days prior to the use of the study drug. In the absence of active autoimmune disease, inhaled or topical steroids and adrenal replacement therapy with prednisone at a dose of ≤ 10 mg per day or equivalent doses of other glucocorticoids are permitted.
* Subjects taking known strong CYP3A4 inhibitors/inducers and P-glycoprotein (P-gp) inhibitors within 14 days prior to the first dose.
* Subjects who have received live virus vaccines (including live attenuated vaccines) within 28 days prior to dosing. Inactivated vaccines are permitted.
* Subjects with a history of psychotropic drug abuse or drug abuse.
* Subjects who have received anti-tumor therapy in the early stage and have not recovered from toxicity (toxicity has not recovered to ≤ Grade 1 according to NCI-CTCAE 5.0). Except for other toxicities (such as alopecia, etc.) that do not affect the safety evaluation of subjects in the opinion of the investigator.
* Subjects with history of other malignancies within 3 years prior to enrollment and not meeting clinical cure criteria. Exceptions are the following: cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the cervix, intraductal carcinoma in situ of the breast, and papillary carcinoma of the thyroid that can be treated locally.
* Subjects with mycosis fungoides, Sézary syndrome, or primary cutaneous T-cell lymphoma.
* Subjects with previous or current central nervous system invasion.
* Subjects with previous or current testicular or breast invasion.
* Subjects with previous or current hemophagocytic syndrome.
* Subjects with previous or current primary or secondary hematologic diseases that may affect bone marrow function in addition to primary malignancies, such as immune thrombocytopenia, autoimmune hemolytic anemia, aplastic anemia, etc.
* Subjects with previous or current acute myeloid leukemia (AML).
* Subjects with previous or current T-cell lymphoblastic lymphoma (T-LBL) or T-lymphoblastic leukemia.
* Subjects who have any history of myeloid malignancy, including myelodysplastic syndrome (MDS), or abnormal tests results of markers related to MDS or myeloproliferative neoplasm (MPN).
* Subjects who previously hadcentral nervous system lesions, or diseases accompanies with central nervous system lesions, including but not limited to, epilepsy, paralysis, stroke, severe brain injury, Alzheimer's disease, Parkinson's disease, cerebellar disease, cerebral organic syndrome, or psychosis, etc.
* Subjects with clinically significant cardiovascular disease.
* Tumor invasion of important peripheral organs and blood vessels (such as heart and pericardium, trachea, esophagus, aorta, superior vena cava, etc.) posing a risk of bleeding or the risk of esophageal tracheal fistula or esophageal pleural fistula.
* Subjects with clinically symptomatic thoracoabdominal effusion or pericardial effusion that are poorly controlled after repeated treatment.
* Subjects with unexplained fever and body temperature>38.0 ℃.
* Subjects who have severe active systemic infection.
* Subjects with a history of tuberculosis infection within one year prior to enrollment, or with a history of active tuberculosis infection more than one year ago without sufficient anti tuberculosis treatment.
* A known history of HIV infection or acquired immunodeficiency syndrome (AIDS), or Anti- Treponema Pallidum test (anti-TP) positive.
* Subjects who have HBV-DNA copy numbers higher than the lower normal limit of the detection value. Subjects with HCV-RNA copy number higher than the lower normal limit of the detection value.
* Subjects who are unable to swallow or has a history of active gastrointestinal inflammation, chronic diarrhea, known diverticular disease, or has undergone gastrectomy or gastric banding that affects drug absorption. But gastroesophageal reflux that has been treated with proton pump inhibitors is allowed (if there is no possibility of drug interaction).
* Subjects with conditions known to have bleeding tendencies, such as von Willebrand disease or hemophilia.
* Subjects who are pregnant or breastfeeding, or expects to conceive within the projected duration of the study.
* Subject who may not be able to complete this study for other reasons or who, in the opinion of the investigator, should not participate the study.

Ages: 18 Days to 70 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) assessed by BICR | 24 mounths

SECONDARY OUTCOMES:
Objective response rate (ORR) | 24 mounths
Time to Response | around 4 months
Duration of response | 24 mounths
Overall survival | around 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No